CLINICAL TRIAL: NCT04182633
Title: Microbiota Transfer Therapy for Children With Autism Spectrum Disorder (ASD) Who Have Gastrointestinal Disorders
Brief Title: MTT for Children With ASD Who Have Gastrointestinal Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEIRB#: 120190306
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Gastro-Intestinal Disorder; Constipation; Diarrhea
Keywords: fecal transplant; fecal microbiota transplant; intestinal microbiota transplant; microbiota transplant; autism; autism spectrum disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Digestive System Diseases; Constipation; Diarrhea; Autistic Disorder | interventions — Vancomycin; polyethylene glycol 3350; Gastrointestinal Microbiome

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized, double-blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Treatment Group (Experimental): This group will receive vancomycin for 14 days, then Miralax for 1 day, then intestinal microbiota for 2 days at high dose, then intestinal microbiota for 12 weeks at a maintenance dose
  Interventions: Combination Product: vancomycin, Miralax, intestinal microbiota
- Group B - Control Group (Miralax only for 1 day) (Placebo Comparator): This group will receive placebo vancomycin for 14 days, then Miralax for 1 day, then placebo intestinal microbiota for 2 days at high dose, then placebo intestinal microbiota for 12 weeks at a maintenance dose
  Interventions: Combination Product: placebo vancomycin, Miralax, placebo intestinal microbiota

INTERVENTIONS:
Combination Product: vancomycin, Miralax, intestinal microbiota — vancomycin for 14 days, then Miralax for 1 day, then intestinal microbiota (high dose for 2 days, then maintenance dose for 12 weeks)
  Arms: Group A - Treatment Group
Combination Product: placebo vancomycin, Miralax, placebo intestinal microbiota — placebo vancomycin for 14 days, then Miralax for 1 day, then placebo intestinal microbiota (high dose for 2 days, then maintenance dose for 12 weeks)
  Arms: Group B - Control Group (Miralax only for 1 day)

SUMMARY:
The investigators propose to investigate Microbiota Transfer Therapy (MTT) for treating children with Autism Spectrum Disorder (ASD) and gastrointestinal problems (primarily constipation and/or diarrhea). MTT involves a combination of 10 days of oral vancomycin (an antibiotic to kill pathogenic bacteria), followed by a bowel cleanse, followed by 12 weeks of Fecal Microbiota (FM).

DETAILED DESCRIPTION:
For children ages 5-17 years with Autism Spectrum Disorder and gastrointestinal problems, a Phase 2 clinical trial will evaluate the safety, tolerability, and efficacy of MTT. The three parts of this trial are described below.

Part 1: Randomized Trial The trial will begin with a randomized, double-blind, placebo-controlled trial which will include a 2-week treatment with oral vancomycin (Group A) or placebo (Group B), then 1 day of Miralax to cleanse the bowel of vancomycin and bacteria/feces (both groups), followed by oral administration of FM (Group A) or placebo (Group B). An initial high dose of FM (or placebo) for two days will be followed by a lower maintenance dose of FM or placebo for 12 weeks.

Part 2: Extension (Group A) and Treatment (Group B)

* For Group A there will be 12-week observation period
* For Group B, there will be treatment similar to that received by the treatment group in Part 1 (partial cross-over, open-label), except that they will not receive vancomycin. So, they will be treated with Miralax followed by an initial high dose of FM for 2 days, and then a maintenance dose of FM for 12 weeks. The purpose of this arm is to determine if vancomycin is necessary or not.

Part 3: Follow-up There will be a follow-up evaluation at 6, 12, and 18 months after treatment ends, to determine long-term safety and efficacy.

Participant duration will be approximately 6.5 months for treatment, and follow-up at 6, 12 and 18 months after treatment ends.

Study duration will be approximately 4 years, including IRB approvals, training staff, recruiting, clinical trial, data analysis, and reporting.

ELIGIBILITY:
Inclusion Criteria for Children with ASD

1. Child aged 5-17 years
2. Diagnosis of autism per the Childhood Autism Rating Scale 2 (CARS-2) and either the Autism Diagnostic Interview-Revised (ADI-R) or the Autism Diagnostic Observation Schedule 2 (ADOS 2).
3. GI disorder as defined below that has lasted for at least 3 years.
4. No changes in medications, supplements, diet, therapies, or education in last 3 months, and no intention to change them during the clinical trial.
5. General good physical health aside from gastrointestinal problems
6. Ability to swallow pills (without chewing)

Exclusion Criteria for Children with ASD

1. Antibiotics in last 3 months (does not apply to topical antibiotics)
2. Probiotics in last 2 months, or fecal transplant in last 12 months
3. Single-gene disorder (Fragile X, etc.)
4. Major brain malformation
5. Tube feeding
6. Severe gastrointestinal problems that require immediate treatment (life-threatening)
7. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions
8. Severely underweight/malnourished (per physician clinical judgement)
9. Unstable, poor health; seizure disorder that is not responsive to treatment or not on stable management or complex type; or other health conditions that would significantly increase their risk of adverse effects (per physician clinical judgement)
10. Recent or scheduled surgeries
11. Current participation in other clinical trials
12. Females who are pregnant or who are sexually active without effective birth control.
13. Allergy or intolerance to vancomycin or Miralax
14. Clinically significant abnormalities at baseline on two blood safety tests: Comprehensive Metabolic Panel and Complete Blood Count with Differential.
15. Psychotropic medication daily use - Current or within past 2 months - which are known to interfere in gastrointestinal function
16. Evidence of significant impairment of immune system, or taking medications that can compromise the immune system, and thus increase risk if exposed to multiple-drug resistant bacteria.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | change in score from baseline to 14 weeks (end of treatment)
  An evaluation by a trained evaluator of autism symptoms. The range is 15-60, and scores in the range of 27-30 or higher are indicative of autism.
Gastrointestinal Symptom Severity Scale (GSRS) | change in score from baseline to 14 weeks (end of treatment)
  A 15-item questionnaire for evaluation of GI symptoms, with each item rated on a scale of 1 (no symptoms) to 7 (severe symptoms), with an average score of 1-7.

SECONDARY OUTCOMES:
Daily Stool Record | change in % abnormal days from baseline (for 2 weeks) vs. week 14 (2 weeks from week 13-14)]
  The DSR is a daily record of bowel movements including Bristol Stool Form scale. It is rated as the % of days with an abnormal report (abnormal stool, no stool, or the use of a gastrointestinal treatment). A higher percentage indicates worse symptoms.
Social Responsiveness Scale 2 | change in score from baseline to 14 weeks (end of treatment)
  A questionnaire about social skills, where higher scores suggest more severe autism. Scores range from 0 to 195, with higher scores indicating more severe problems.
Aberrant Behavior Checklist | change in score from baseline to 14 weeks (end of treatment)
  A questionnaire about aberrant behaviors. Scores range from 0 to 174, with higher scores indicating more severe behaviors

CONTACTS AND LOCATIONS:
Overall Officials: James B Adams, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The web page for the research group leading this study — http://autism.asu.edu